CLINICAL TRIAL: NCT03898544
Title: Assessment at Short Term of the Gait Kinematics After Primary TKA (Stryker) Versus After Revision TKA. Prospective and Controlled Study.
Brief Title: Gait Kinematics After Primary Total Knee Arthroplasty (TKA) Versus Revision TKA
Acronym: Stryker-KneeKG
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Stryker Nordic (Industry)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0089; 2019-A00478-49 (Other: ANSM)
Record Dates: First submitted 2019-03-29; First posted 2019-04-02 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Knee Arthroplasty, Total; Gait Analysis
Keywords: gait kinematics; TKA
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group primary TKA: Patients operated of primary TKA Stryker for knee osteoarthritis.
  Interventions: Device: Group primary TKA
- Group TKA revision: Patients operated of a first revision of TKA for a mechanical failure, with the revision Stryker TKA
  Interventions: Device: Group TKA revision

INTERVENTIONS:
Device: Group primary TKA — Assessment by gait kinematics analysis The total knee arthroplasty will be performed as usual with the dedicated instrumentation.
  The gait kinematics analysis will be performed with the KneeKG system on a treadmill, with infrared sensors (IR) on the leg. This system is not invasive. The IR sensors are positioned on the pelvis, the distal femur and the tibial crest. This system records the flexion/extension, the varus/valgus and the rotation during the walking (1 minute of walking).
  Other Names: Total knee arthroplasty
  Groups: Group primary TKA
Device: Group TKA revision — Assessment by gait kinematics analysis The total knee arthroplasty will be performed as usual with the dedicated instrumentation.
  The gait kinematics analysis will be performed with the KneeKG system on a treadmill, with infrared sensors on the leg. This system is not invasive. The IR sensors are positioned on the pelvis, the distal femur and the tibial crest. This system records the flexion/extension, the varus/valgus and the rotation during the walking (1 minute of walking).
  Other Names: Total knee arthroplasty
  Groups: Group TKA revision

SUMMARY:
The functional outcomes after TKA are satisfying with a full recovery at 6 months - 1 year. Nevertheless, the revisions of TKA have often lower functional results than primary TKA with a long delay of recovery. The Stryker TKA present the same device for primary TKA and for revision.

The aim of this study is to compare the gait kinematics at 6 months after primary Stryker TKA or Revision Stryker TKA to assess if the objective outcomes are similar with this device.

ELIGIBILITY:
Inclusion Criteria:

* Primary TKA group: symptomatic femorotibial osteoarthritis, with an indication of primary TKA (as Triathlon Stryker)
* Revision group: first TKA removal in 1 step for mechanical failure, by a revision TKA (as Triathlon Stryker)

Exclusion Criteria:

* Septic failure
* Second or more failure in the revision group
* Associated surgical procedure as osteotomy, allograft…
* Not full weight bearing postoperatively
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary TKA group: symptomatic femorotibial osteoarthritis, with an indication of primary TKA (as Triathlon Stryker)
  Revision group: first TKA removal in 1 step for mechanical failure, by a revision TKA (as Triathlon Stryker)
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Femorotibial mechanical axis (varus, valgus) analysis | at 6 months postoperatively
  These parameters are measured with the KneeKG system during the walking
range of motion (flexion, extension) analysis | at 6 months postoperatively
  These parameters are measured with the KneeKG system during the walking
internal/external rotation analysis | at 6 months postoperatively
  These parameter is measured with the KneeKG system during the walking
Walking speed | at 6 months postoperatively
  These parameter is measured with the KneeKG system

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Lustig, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital de la Croix Rousse, Lyon, France